CLINICAL TRIAL: NCT02938871
Title: Effect of Synbiotic on Postoperative Complications After Liver Transplantation - A Randomized Double-blind Clinical Trial
Brief Title: Effect of Synbiotic on Postoperative Complications After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 160012
Record Dates: First submitted 2016-10-07; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Liver Disease
Keywords: synbiotic; infections; probiotics; liver transplantation
MeSH Terms: conditions — Liver Diseases; Infections | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synbiotic (Active Comparator): The patients of this group will receive 6 grams of synbiotic composition, to be administered via feeding tube or orally, twice time a day, for 15 consecutive days.
  Interventions: Dietary Supplement: Synbiotic
- Control (Placebo Comparator): The patients of this group will receive 6 grams of maltodextrin, to be administered via feeding tube or orally, twice time a day, for 15 consecutive days.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Synbiotic — The patients of this group will receive 6 grams of synbiotic composition, to be administered via feeding tube or orally, twice time a day, for 15 consecutive days.
  Arms: Synbiotic
Dietary Supplement: Control — The patients of this group will receive 6 grams of maltodextrin, to be administered via feeding tube or orally, twice time a day, for 15 consecutive days.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the use of synbiotic in patients after liver transplantation and assess the effect of these agents on postoperative infections, antibiotic use, length of hospital stay, mortality and nutritional status.

DETAILED DESCRIPTION:
All patients who are undergoing liver transplantation at the Hospital de Clinicas de Porto Alegre over the next 18 months will be informed of the purpose of the study. The patients or their legal guardians provided will written an informed consent for participation at the study.

The patients will be allocated to the intervention or control groups by randomization in blocks. The intervention group will receive a synbiotic composition (Lactobacillus acidophilus NCFM SD5221 10bilhões; Lactobacillus rhamnosus HN001 5675 SD 10 billion; Lactobacillus paracasei LPC SD 5275 - 37 10 billion; Bifidobacterium lactis SD 5674 HN0019 10 billion; Fructooligosaccharide 5.5 g) and the control group will receive 6 g of maltodextrin.The patients will received a synbiotic composition or maltodextrin for 15 days, twice times a day, after liver transplantation, when the patients are able to start feeding.

Patients will be evaluated for the occurrence of infections, need for additional antibiotics, length of hospital stay and mortality.

The Nutritional assessment will be carried out before and after surgery. All information will be collected and stored prospectively and the clinical trial will follow the instructions of the Consolidated Standards of Reporting Trials - CONSORT 2010.

ELIGIBILITY:
Inclusion Criteria:

* All adults patients who are undergoing liver transplantation

Exclusion Criteria:

* patients on parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of synbiotic on postoperative infection after liver transplantation | 15 days
  positive blood culture

SECONDARY OUTCOMES:
Identify length of postoperative hospital stay | up to 12 weeks
  length of hospital stay will be counted in days
Identify duration of antibiotic therapy | up to 30 days
  The duration of antibiotic therapy will be counted in days
Identify mortality | up to 30 days
  It will be considered mortality the events occurring up to 30 days after surgery
Identify nutritional status of patients undergoing liver transplantation using the questionnaire of subjective global assessment and the global nutritional assessment proposed by Royal Free Hospital | until one month before surgery and 10 days after surgery

OTHER OUTCOMES:
Identify nutritional status of patients undergoing liver transplantation using the measurement of non-dominant handgrip and the measurement of adductor polices muscle | until one month before surgery and 10 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Cleber Kruel, Doctor, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cooper TE, Scholes-Robertson N, Craig JC, Hawley CM, Howell M, Johnson DW, Teixeira-Pinto A, Jaure A, Wong G. Synbiotics, prebiotics and probiotics for solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 20;9(9):CD014804. doi: 10.1002/14651858.CD014804.pub2. PMID 36126902